CLINICAL TRIAL: NCT00373295
Title: Effect of Baclofen on Marijuana Withdrawal and Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 5232; 5P50DA009236 (NIH)
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Marijuana Dependence
Keywords: Baclofen; Marijuana Dependence; Marijuana Withdrawal
MeSH Terms: conditions — Marijuana Abuse | interventions — Baclofen; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Baclofen 60 mg, Placebo, Baclofen 90 mg (Experimental): Baclofen (60mg/day or 90 mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (0, 20, 30mg) were administered 3 times per day (0900, 1530, 2200).
  Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Baclofen; Drug: Marijuana; Drug: Placebo
- Baclofen 90 mg, Placebo, Baclofen 60 mg (Experimental): Baclofen (60mg/day or 90 mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (0, 20, 30mg) were administered 3 times per day (0900, 1530, 2200).
  Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Baclofen; Drug: Marijuana; Drug: Placebo
- Baclofen 60 mg, Baclofen 90 mg, Placebo (Experimental): Baclofen (60mg/day or 90 mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (0, 20, 30mg) were administered 3 times per day (0900, 1530, 2200).
  Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Baclofen; Drug: Marijuana; Drug: Placebo
- Baclofen 90 mg, Baclofen 60 mg, Placebo (Experimental): Baclofen (60mg/day or 90 mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (0, 20, 30mg) were administered 3 times per day (0900, 1530, 2200).
  Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Baclofen; Drug: Marijuana; Drug: Placebo
- Placebo, Baclofen 90 mg, Baclofen 60 mg (Experimental): Baclofen (60mg/day or 90 mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (0, 20, 30mg) were administered 3 times per day (0900, 1530, 2200).
  Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Baclofen; Drug: Marijuana; Drug: Placebo
- Placebo, Baclofen 60 mg, Baclofen 90 mg (Experimental): Baclofen (60mg/day or 90 mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (0, 20, 30mg) were administered 3 times per day (0900, 1530, 2200).
  Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Interventions: Drug: Baclofen; Drug: Marijuana; Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Baclofen (60mg/day or 90 mg/day): Packaged medication in size 00 opaque capsules with riboflavin filler. Study capsules (0, 20, 30mg) were administered 3 times per day (0900, 1530, 2200).
  Other Names: Lioresal
Drug: Marijuana — Marijuana: Participants each received a single marijuana cigarette (provided by the National Institute on Drug Abuse) at each smoking occasion. Marijuana cigarettes were stored frozen in an airtight container and humidified at room temperature for 24 h prior to use.
  Other Names: cannabis
Drug: Placebo

SUMMARY:
The purpose of this study is to determine if baclofen dose-dependently decreases marijuana's direct effects and symptoms of marijuana withdrawal and thus decreases marijuana relapse.

DETAILED DESCRIPTION:
Only a small percentage of dependent-marijuana smokers who are seeking treatment for their marijuana use are able to achieve sustained abstinence. The objective of this study is to investigate the interaction between marijuana and the potential treatment medication, baclofen, with the direct goal of using this information to improve marijuana treatment outcome. GABAB agonists such as baclofen have been shown to attenuate the self-administration of cocaine, heroin, alcohol and nicotine (see Cousins et al., 2002; Haney et al., 2006). Baclofen also appears to decrease withdrawal symptoms in heroin and alcohol abusers (Akhondzadeh et al., 2000; Addolorato et al., 2000). The purpose of this study is to determine if baclofen dose-dependently decreases marijuana's direct effects and symptoms of marijuana withdrawal and thus decreases marijuana relapse in our laboratory model. For the purposes of this model, relapse is defined as a return to marijuana use after a period of abstinence. The study will utilize an inpatient/outpatient, counter-balanced design, with each participant maintained on each of three medication conditions for 16 days: placebo and baclofen (60, 90 mg/day). Participants will begin taking capsules during the outpatient phase so that the dose can be incremented up to the maintenance dose prior to the first inpatient day. Further, clinical studies have shown that baclofen is most effective at decreasing cocaine's effects when administered for several weeks. During the inpatient study phases, participants will have the opportunity to self-administer placebo or active marijuana 6 times per day. This study will provide important information of the effect of baclofen as a potential treatment medication for marijuana dependence.

ELIGIBILITY:
Inclusion Criteria:

* Current marijuana use: average of 3 marijuana cigarettes at least 4 times per week for the past 4 weeks
* Able to perform study procedures
* 21-45 years of age
* Women practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD)

Exclusion Criteria:

* Current, repeated illicit drug use (other than marijuana)
* Presence of significant medical illness(e.g., diabetes, cardiovascular disease, hypertension, examination, laboratory clinically significant laboratory abnormalities)
* History of heart disease
* Request for drug treatment
* Current parole or probation
* Pregnancy or current lactation
* Recent history of significant violent behavior
* Major current Axis I psychopathology(e.g., major depressive disorder, bipolar disorder, suicide risk, schizophrenia)
* Current use of any prescription or over-the-counter medication

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Haney M, Hart CL, Vosburg SK, Comer SD, Reed SC, Cooper ZD, Foltin RW. Effects of baclofen and mirtazapine on a laboratory model of marijuana withdrawal and relapse. Psychopharmacology (Berl). 2010 Aug;211(2):233-44. doi: 10.1007/s00213-010-1888-6. Epub 2010 Jun 3. PMID 20521030

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 participants were enrolled, but 10 participants were randomized. Three volunteers (1 female, 2 male) dropped out of the study during the marijuana abstinence phase (two were on baclofen and one was on placebo).
Groups:
- Baclofen 60 mg, Placebo, Baclofen 90 mg: participants received baclofen (60 mg/day) for 8 days, followed by placebo for 8 days, then baclofen (90mg/day) for 8 days.
- Baclofen 90 mg, Placebo, Baclofen 60 mg: participants received baclofen (90mg/day) for 8 days, followed by placebo for 8 days, then baclofen (60mg/day) for 8 days.
- Baclofen 60 mg, Baclofen 90 mg, Placebo: participants received baclofen (60mg/day) for 8 days, followed by baclofen (90mg/day) for 8 days, then placebo for 8 days.
- Baclofen 90 mg, Baclofen 60 mg, Placebo: participants received baclofen (90mg/day) for 8 days, followed by baclofen (60mg/day) for 8 days, and then placebo for 8 days.
- Placebo, Baclofen 90 mg, Baclofen 60 mg: participants received placebo for 8 days, followed by baclofen (90mg/day) for 8 days, then baclofen (60mg/day) for 8 days.
- Placebo, Baclofen 60 mg, Baclofen 90 mg: participants received placebo for 8 days, followed by baclofen (60mg/day) for 8 days, then baclofen (90mg/day) for 8 days.
Period: Intervention 1 (8 Days)
Arm/Group | Baclofen 60 mg, Placebo, Baclofen 90 mg | Baclofen 90 mg, Placebo, Baclofen 60 mg | Baclofen 60 mg, Baclofen 90 mg, Placebo | Baclofen 90 mg, Baclofen 60 mg, Placebo | Placebo, Baclofen 90 mg, Baclofen 60 mg | Placebo, Baclofen 60 mg, Baclofen 90 mg
Started | 2 | 3 | 1 | 2 | 3 | 2
Completed | 2 | 1 | 1 | 2 | 2 | 2
Not Completed | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 1 | 0
Period: Intervention 2 (8 Days)
Arm/Group | Baclofen 60 mg, Placebo, Baclofen 90 mg | Baclofen 90 mg, Placebo, Baclofen 60 mg | Baclofen 60 mg, Baclofen 90 mg, Placebo | Baclofen 90 mg, Baclofen 60 mg, Placebo | Placebo, Baclofen 90 mg, Baclofen 60 mg | Placebo, Baclofen 60 mg, Baclofen 90 mg
Started | 2 | 1 | 1 | 2 | 2 | 2
Completed | 2 | 1 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3 (8 Days)
Arm/Group | Baclofen 60 mg, Placebo, Baclofen 90 mg | Baclofen 90 mg, Placebo, Baclofen 60 mg | Baclofen 60 mg, Baclofen 90 mg, Placebo | Baclofen 90 mg, Baclofen 60 mg, Placebo | Placebo, Baclofen 90 mg, Baclofen 60 mg | Placebo, Baclofen 60 mg, Baclofen 90 mg
Started | 2 | 1 | 1 | 2 | 2 | 2
Completed | 2 | 1 | 1 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants received placebo, baclofen (60mg) and baclofen (90mg) and smoked Marijuana (5.3% THC).
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Measure of Relapse: Change in Money Spent Between Baseline and Relapse Phase
Description: This is a measure of marijuana self-administration and relapse since each initial puff costs $7 and is a burden to overcome just to smoke.
  Over each 3 day period, the puffs chosen by each participant is averaged for a single value.
Time Frame: Days 1-3 (Baseline) and Days 6-8 (Relapse Phase)
Measure: Mean (Standard Deviation); unit: dollars spent on marijuana
Groups:
- Baclofen 60, Marijuana: baclofen (60 mg)/day
  Baclofen: measured baclofen's effects on marijuana withdrawal and relapse relative to placebo
  Marijuana: measured baclofen's effects on marijuana withdrawal and relapse
- Baclofen 90, Marijuana: baclofen (90 mg)/day
  Baclofen: measured baclofen's effects on marijuana withdrawal and relapse relative to placebo
  Marijuana: measured baclofen's effects on marijuana withdrawal and relapse
Arm/Group | Baclofen 60, Marijuana | Placebo, Marijuana | Baclofen 90, Marijuana
Number analyzed (Participants) | 13 | 13 | 13
dollars spent on marijuana | 7.15 (1.85) | 9.77 (2.30) | 7.25 (2.10)

ADVERSE EVENTS:
Groups:
- Placebo, Marijuana: Marijuana: measured baclofen's effects on marijuana withdrawal and relapse
Arm/Group | Baclofen 60, Marijuana | Baclofen 90, Marijuana | Placebo, Marijuana
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 2/13 | 0/13 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen 60, Marijuana (N=13) | Baclofen 90, Marijuana (N=13) | Placebo, Marijuana (N=13)
mild headache (Social circumstances) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No